CLINICAL TRIAL: NCT03677011
Title: Andrositol® TEST as Diagnostic Assay to Predict the Fertilization Potential of the Sperm in the in Vitro Fertilization (IVF) Procedures.
Brief Title: Andrositol® TEST as Diagnostic Assay to Predict the Fertilization Potential in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 100006555
Record Dates: First submitted 2018-07-25; First posted 2018-09-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Male Infertility
Keywords: myo-inositol; fertilization rate; infertility; Intracytoplasmic Sperm Injection; sperm
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- category 1 (Other): Low responder
  Interventions: Diagnostic Test: Andrositol® Test
- category 2 (Other): Medium Responder and High Responder
  Interventions: Diagnostic Test: Andrositol® Test

INTERVENTIONS:
Diagnostic Test: Andrositol® Test — The intervention consists in the addiction of myo-inositol directly to the semen identifying the quality of sperm prior ICSI procedure

SUMMARY:
Andrositol® test allows to obtain additional information besides the WHO parameters and to evaluate the semen energetic status. The diagnosis is performed by analyzing the semen at two different time points: before the treatment and 30' after the addiction of myo-inositol directly to the semen. The purpose of this study is to evaluate if the responsiveness to the Andrositol® test of a sperm sample can be predictive of its fertilization rate in an ICSI (Intracytoplasmic Sperm Injection) cycle (primary outcome). Secondary outcomes as embryo development, embryo euploidy status and embryo implantation rate will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male partners of couples undergoing an egg donor cycles

Exclusion Criteria:

* sperm volume lower than 1 ml
* sperm count lower than 5 X 106 /ml
* total sperm motility lower than 10%

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since we are testing the predictive value of a sperm test, the gender of the prospective subjects will be restricted to male partners of couples undergoing an ICSI treatment.
Enrollment: 249 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
increment of the fertilization rate | up to 20 hours after ICSI
  measurement of the % oocytes become fertilized by sperm cells. This outcome, is calculated for each patient at day + 1 (14-20h after icsi)

SECONDARY OUTCOMES:
Increment of implantation rate | up to 10 days after ICSI
  implantation rate is calculated as the number of gestational sacs observed at echographic screening at +5 weeks of pregnancy divided by the number of embryos transferred
embryo development | up to 6 days after ICSI
  the number of blastocysts for each patient at day +5, +6, +7
embryo euploidy | from 10 days after ICSI
  Embryo euploidy for each patient at day +10

CONTACTS AND LOCATIONS:
Overall Officials: Tih T. Tan, Ms, Principal Investigator — HRC Pasadena 333 S Arroyo Pkwy Fl 3 Pasadena, CA 91105
Locations (1):
- HRC Pasadena, Pasadena, California, United States